CLINICAL TRIAL: NCT06966453
Title: A Phase 1b/2, Open-Label, Multicohort Study of Disitamab Vedotin in Adults With HER2 Expressing Advanced Breast Cancer
Brief Title: A Study of Disitamab Vedotin in Adults With HER2 Expressing Advanced Breast Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C5731006; 2025-521003-52-00 (EU CTIS Number); SGNDV-006 (Other: Seagen)
Record Dates: First submitted 2025-05-09; First posted 2025-05-11 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer; Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — disitamab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1: HER2+ locally advanced or metastatic breast cancer (Experimental): disitamab vedotin monotherapy
  Interventions: Drug: Disitamab vedotin
- Cohort 2: HR+, HER2-low locally advanced or metastatic breast cancer (Experimental): disitamab vedotin monotherapy
  Interventions: Drug: Disitamab vedotin
- Cohort 3: HR+, HER2 ultra-low or HR-negative, HER2-low locally advanced or metastatic breast cancer (Experimental): disitamab vedotin monotherapy
  Interventions: Drug: Disitamab vedotin

INTERVENTIONS:
Drug: Disitamab vedotin — Given into the vein (IV; intravenous) every 2 weeks.
  Other Names: RC48; RC48-ADC

SUMMARY:
The purpose of this clinical study is to learn about the safety and effects of the study medicine (called disitamab vedotin) for the possible treatment of people with breast cancer that is hard to treat and has spread in the body (advanced cancer).

This study is seeking participants who:

* have breast cancer that is hard to treat and has spread in the body (advanced cancer)
* have tumors that have HER2 on them
* have received previous treatment for their advanced breast cancer

All participants in this study will receive disitamab vedotin at the study clinic once every 2 weeks as an intravenous (IV) infusion (given directly into a vein).

Participants will take the study medicine until they or their doctor decides to stop. This might be because their cancer is getting worse, the study medicine is no longer helping, they have bad side effects, or they wish to stop taking the study medicine. During this time, the participants will have study visits every 2 weeks. After the participants have stopped taking the study medicine, they will have follow-up visits about every 6 weeks unless their cancer gets worse. After that, they will have follow-up phone calls about every 12 weeks.

The study team will look at the experiences of people receiving the study medicine. This will help the study team decide if the study medicine is safe and effective.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed diagnosis of locally-advanced, unresectable, or metastatic breast carcinoma.
* Human epidermal growth factor receptor 2 (HER2) and hormone receptor (HR) status appropriate for enrollment in cohort.
* HER2 status determined by most recent local assessment based on American Society of Clinical Oncology (ASCO) and College of American Pathologists (CAP) guidelines for assessment of HER2 in BC for interpretation of HER2 expression and amplification
* HER2+: immunohistochemistry (IHC) 3+ or IHC 2+/in situ hybridization (ISH)+
* HER2-low: IHC 1+/ISH-negative or untested or IHC 2+/ISH-negative
* HER2-ultralow: IHC 0 with membrane staining (any staining of the membrane in >0 and ≤10% of cancer cells) o HR+ disease is determined as either estrogen receptor (ER) and/or progesterone receptor (PgR) positive [ER or PgR ≥1%]) and HR negative disease is determined as both ER and PR negative [ER and PgR <1%]) per ASCO/CAP guidelines in the advanced disease setting. If a patient has had multiple ER/PgR results for advanced disease, the most recent test result will be used to confirm eligibility.

Prior therapy requirements for Cohort 1 (HER2+, HR+ or HR- participants):

* Received prior trastuzumab, pertuzumab and a taxane if available as local first line standard of care therapy for advanced disease.
* Prior tucatinib based therapy is allowed.
* Must have progression on or after, or be intolerant to, T-DXd in any line advanced disease setting.
* No more than 3 prior systemic cytotoxic therapy regimens (including antibody drug conjugates [ADCs]) for Locally Advanced (LA)/metastatic breast cancer (mBC). Participants previously treated with (neo)adjuvant cytotoxic therapy and have disease relapsed within 6 months of cytotoxic treatment is considered to have received 1 line of cytotoxic therapy for LA/mBC.

Prior therapy requirements for Cohort 2 (HR+/HER2-low participants):

* No more than 3 prior systemic cytotoxic therapy regimens (including ADCs) for LA/mBC. Participants previously treated with (neo)adjuvant cytotoxic therapy and have disease relapsed within 6 months of cytotoxic treatment is considered to have received 1 line of cytotoxic therapy for LA/mBC.
* Participants with known germline breast cancer gene (BRCA) mutation must have received a poly-ADP ribose polymerase (PARP) inhibitor, where available and not medically contraindicated.
* Must have progression on or after, or be intolerant to, trastuzumab deruxtecan (T-DXd) in any line advanced disease setting.
* Must have intolerance to endocrine therapy (ET) or ET refractory disease:
* Progressed on ≥2 lines of ET for LA/mBC AND had received a cyclin-dependent kinase (CDK)4/6 inhibitor in the adjuvant or metastatic setting if available as local standard of care and not contraindicated.

OR

• Progressed on 1 line of ET for LA/mBC AND had a relapse while on adjuvant ET after definitive surgery for primary tumor AND had received a cyclin-dependent kinase (CDK) 4/6 inhibitor in the adjuvant or advanced setting if available as local standard of care and not contraindicated.

Prior therapy requirements for Cohort 3 (HR+/HER2-ultralow or HR-/HER2-low [HER2 low TNBC] participants):

* No more than 4 prior systemic cytotoxic chemotherapy regimens (including ADCs) for advanced or mBC. Participants previously treated with (neo)adjuvant cytotoxic therapy and have disease relapsed within 6 months of cytotoxic treatment is considered to have received 1 line of cytotoxic therapy for LA/mBC.
* Known germline BRCA mutation must have received a PARP-inhibitor if available as local standard of care therapy and not medically contraindicated.
* Prior sacituzumab govitecan is allowed.
* Prior T-DXd is allowed.
* Participants with HR negative (TNBC), HER2-low and programmed cell death receptor ligand 1 (PD-L1)-positive (combined positive score [CPS] ≥10) tumors must have received pembrolizumab (or other PD-L1 inhibitor) with chemotherapy if available as local standard of care therapy and not medically contraindicated.
* Participants with HR+/HER2-ultra low tumors must have received at least 1 antihormonal therapy in any setting or be ineligible for ET.
* Participants with HR+/HER2-ultra low tumors must have had prior therapy with a CDK4/6 inhibitor in the adjuvant or advanced setting.

Exclusion Criteria

* Known hypersensitivity to any excipient contained in the drug formulation of disitamab vedotin.
* Active central nervous system (CNS) and/or leptomeningeal metastasis.
* Participants with a history of other invasive malignancy within 3 years before the Cycle 1 Day 1 (C1D1) of study intervention, or any evidence of residual disease from a previously diagnosed malignancy.
* Prior therapy with ADCs with MMAE payload.
* Participants who have received prior systemic anticancer treatment or radiotherapy within 2 weeks, or 5 half-lives, whichever is shorter, prior to C1D1 of study intervention. Note: If the last immediate anticancer treatment contained an antibody-based agent(s), then an interval of 28 days or 5 half-lives (whichever is shorter) of the agent(s) prior to receiving the study intervention treatment is required.

  * Participants must have recovered from all adverse events due to previous therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2027-10-25 (Estimated); Study Completion 2030-01-27 (Estimated)

PRIMARY OUTCOMES:
Objective response (OR) by investigator assessment | From Cycle 1 Day 1 until disease progression by investigator assessment per RECIST version 1.1, or death due to any cause, whichever is earlier; up to approximately 2 years
  The primary endpoint OR by investigator assessment is defined as the proportion of participants with confirmed CR or PR as determined by investigator per RECIST Version 1.1.

SECONDARY OUTCOMES:
Duration of response (DOR) per RECIST v1.1 by investigator assessment | From first documentation of objective response (CR or PR) by investigator assessment per RECIST version 1.1 that is subsequently confirmed, to the first documentation of progressive disease or to death due to any cause; up to approximately 2 years
  DOR by investigator assessment is defined as the time from first documentation of objective response (CR or PR) by investigator assessment per RECIST version 1.1 that is subsequently confirmed, to the first documentation of progressive disease or to death due to any cause, whichever comes first.
Disease control rate (DCR) (confirmed CR, confirmed PR, and stable disease) per RECIST v1.1 by investigator assessment | From Cycle 1 Day 1 until disease progression by investigator assessment per RECIST version 1.1, or death due to any cause, whichever is earlier; up to approximately 2 years
  DCR by investigator assessment is defined as the proportion of participants with CR or PR with confirmation, or Stable Disease (SD) by investigator assessment per RECIST version 1.1.
Progression-free survival (PFS) per RECIST v1.1 by investigator assessment | From Cycle 1 Day 1 until disease progression by investigator assessment per RECIST version 1.1, or death due to any cause, whichever is earlier; ; up to approximately 2 years
  PFS by investigator assessment is defined as the time from C1D1 to the first documentation of disease progression as determined by investigator per RECIST version 1.1, or to death due to any cause, whichever comes first.
Overall survival (OS) | From Cycle 1 Day 1 until death due to any cause; up to approximately 3 years
  OS is defined as the time from C1D1 to date of death due to any cause.
PK Parameter: Serum Concentrations of disitamab vedotin, total antibody, and unconjugated MMAE | From Cycle 1 Day 1 to end of treatment; up to approximately 2 years
  The Antibody-drug conjugate (TAb), and unconjugated Monomethyl auristatin E (MMAE) concentrations for disitamab vedotin summarized at each PK sampling time point.
Incidence of anti-drug antibodies (ADA) against disitamab vedotin | From Cycle 1 Day 1 to end of treatment; up to approximately 2 years
  The percentage of participants with positive ADA will be summarized.
Incidence of Adverse Events (AE) and Serious Adverse Events (SAE) | Up to approximately 2 years
  Type, incidence, severity, seriousness, and relatedness of AEs. Type, incidence, and severity of laboratory abnormalities and significant changes from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (97):
- United States (88):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Southern Cancer Center, PC, Foley, Alabama
  - Southern Cancer Center, PC, Mobile, Alabama
  - Los Angeles Cancer Network, Fountain Valley, California
  - Los Angeles Hematology Oncology Medical Group, Glendale, California
  - Los Angeles Cancer Network, Los Angeles, California
  - Valkyrie Clinical Trials, Los Angeles, California
  - Mission Community Hospital (Satellite Site), Los Angeles, California
  - Clinical and Translational Research Unit (CTRU), Palo Alto, California
  - Stanford Cancer Center, Palo Alto, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Stanford Health Care, Investigational Drug Service, Stanford, California
  - Los Angeles Hematology Oncology Medical Group, Van Nuys, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Boulder, Colorado
  - Rocky Mountain Cancer Centers, LLP, Centennial, Colorado
  - Rocky Mountain Cancer Centers, LLP, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP, Englewood, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, LLP, Littleton, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, LLP, Longmont, Colorado
  - Rocky Mountain Cancer Centers, LLP, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, LLP, Thornton, Colorado
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Lecanto, Florida
  - Florida Cancer Specialists, Ocala, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tallahassee, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, The Villages, Florida
  - Florida Cancer Specialists, Trinity, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - Florida Cancer Specialists, Winter Park, Florida
  - Oncology Associates of Oregon, P.C., Albany, Oregon
  - Oncology Associates of Oregon, P.C., Corvallis, Oregon
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Oncology Associates of Oregon, P.C., Springfield, Oregon
  - Alliance Cancer Specialists, PC, Bensalem, Pennsylvania
  - Alliance Cancer Specialists, PC, Doylestown, Pennsylvania
  - Alliance Cancer Specialists, PC, Horsham, Pennsylvania
  - Alliance Cancer Specialists, PC, Langhorne, Pennsylvania
  - Alliance Cancer Specialists, PC, Media, Pennsylvania
  - Alliance Cancer Specialists, PC, Sellersville, Pennsylvania
  - Alliance Cancer Specialists, PC, Wynnewood, Pennsylvania
  - Sarah Cannon Research Institute - Pharmacy, Nashville, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology-Northeast Texas, Allen, Texas
  - Texas Oncology - DFW, Arlington, Texas
  - Texas Oncology - DFW, Bedford, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Texas Oncology-Northeast Texas, Denison, Texas
  - Texas Oncology-Northeast Texas, Denton, Texas
  - Texas Oncology-Northeast Texas, Flower Mound, Texas
  - Texas Oncology - DFW, Fort Worth, Texas
  - Texas Oncology - DFW, Grapevine, Texas
  - US Oncology Investigation Products Center(IPC), Irving, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - Texas Oncology-Northeast Texas, Lewisville, Texas
  - Texas Oncology-Northeast Texas, Longview, Texas
  - Texas Oncology-Northeast Texas, McKinney, Texas
  - Texas Oncology-Northeast Texas, Palestine, Texas
  - Texas Oncology - Northeast Texas, Paris, Texas
  - Texas Oncology-Northeast Texas, Paris, Texas
  - Texas Oncology - DFW, Plano, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Virginia Cancer Specialists, PC, Arlington, Virginia
  - Oncology & Hematology Associates of Southwest Virginia Inc dba Blue Ridge Cancer Care, Blacksburg, Virginia
  - Virginia Oncology Associates, Chesapeake, Virginia
  - Virginia Cancer Specialists, PC, Fairfax, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Low Moor, Virginia
  - Virginia Cancer Specialists, PC, Manassas, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Specialists, PC, Reston, Virginia
  - Oncology & Hematology Associates of Southwest Virginia Inc dba Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology & Hematology Associates of Southwest Virginia Inc dba Blue Ridge Cancer Care, Salem, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
  - Virginia Oncology Associates, Williamsburg, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Wytheville, Virginia
- Australia (4):
  - Blacktown Hospital, Blacktown, New South Wales
  - Royal Brisbane and Women's Hospital, Brisbane, Queensland
  - Metro North Hospital and Health Service, Herston, Queensland
  - Western Health-Sunshine & Footscray Hospitals, St Albans, Victoria
- Canada (2):
  - Waterloo Regional Health Network, Kitchener, Ontario
  - Lakeridge Health, Oshawa, Ontario
- Japan (2):
  - Osaka University Hospital, Suita, Osaka
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
- Pan American Center for Oncology Trials, LLC, Rio Piedras, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5731006